CLINICAL TRIAL: NCT03965910
Title: Demonstration the Importance of the Early Rehabilitation in Stroke Patients Based on Diffüsion Tensor Imaging Data
Brief Title: Importance of Early Rehabilitation in Stroke Patients
Acronym: stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Yaşar Keskin, Principal Investigator at Department of Physical Medicine and Rehabilitation at Bezmialem Vakif University, Medical Doctor, Bezmialem Vakif University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28/09/2016-12 /25
Record Dates: First submitted 2019-04-10; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; diffusion tensor imaging
MeSH Terms: conditions — Stroke | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The clinician evaluating the patient and the radiologist evaluating the MRI were blinded to the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Other): Group 1:Early rehabilitation
  Interventions: Other: Demonstration the Importance of Early Rehabilitation in Stroke Patients Based on Diffusion Tensor Imaging Data
- group 2 (Other): Group 2:Late rehabilitation
  Interventions: Other: Demonstration the Importance of Early Rehabilitation in Stroke Patients Based on Diffusion Tensor Imaging Data

INTERVENTIONS:
Other: Demonstration the Importance of Early Rehabilitation in Stroke Patients Based on Diffusion Tensor Imaging Data — Twenty-eight stroke patients aged 36-72 years admitted to the our Physical Medicine and Rehabilitation Outpatient Clinics were included in this prospective study. After the approval of the ethics committee, written informed consent was obtained from the patients after they were informed about the content and purpose of the study, the schedule of rehabilitation to be administered, and the features of cranial magnetic resonance imaging (MRI) to be performed. Patients with confirmed diagnosis of stroke by computed tomography and/or MRI techniques were randomized into two groups according to the onset of post-stroke rehabilitation. The patients were randomized according to the duration of their admission to our clinic for rehabilitation. Group 1 consisted of patients admitted to our clinic within 1-4 weeks after stroke; Group 2 consisted of patients admitted within 5-8 weeks after stroke.
  Late initiation of rehabilitation in Group 2 patients is not a condition related to our clinic.
  Other Names: Poststroke rehabilitation and diffusion tensor imaging

SUMMARY:
Stroke is one of the leading health problems in the community and it is the most common life-threatening neurological disease impairing the quality of life. Early rehabilitation of stroke is very important. The purpose of our study was to evaluate, through clinical examination, whether there was any difference between patients who underwent early rehabilitation and those who underwent late rehabilitation in terms of improvements in motor and functional impairment after rehabilitation, and also to evaluate this difference objectively by analyzing white-matter pathways (corticospinal tracts) using DTI.

DETAILED DESCRIPTION:
Methods: Twenty-eight (28) adults (12 women, 16 men, average age 58 years) with first-time stroke who met the study criteria were divided into two groups depending on the duration of their stroke at the time of their presentation to our facility. Group 1 consisted of patients who underwent rehabilitation program within the first 1-4 weeks after stroke, whereas Group 2 consisted of patients who underwent rehabilitation program within 5-8 weeks after stroke. Both groups were evaluated using the BRS, FMA scale, FAC and BI scales. For cranial imaging, DTI was obtained 1 day before and 1 day after treatment. FA and ADC values of corticospinal tracts were performed using DTI.

Intervention: Patients were enrolled in a rehabilitation program, which was designed for a total of 4 weeks, with daily sessions lasting a total of 1 h on 5 days of a week.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering cerebrovascular accident (CVA)-associated stroke for the first time with a cortical or subcortical unilateral ischemia or hemorrhage
* The patients aged 35-75 years
* Patiients with ability to understand and follow the instructions
* Patients with the absence of serious cognitive deficits.

Exclusion Criteria:

* Patients who had spinal-cord lesion
* Patients who had history of traumatic brain injury,
* Patients who had accompanying neurological disease (multiple sclerosis, Parkinson's disease, dementia)
* Patients who had tumor
* Patients who had history of convulsions

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in Cranial diffusion tractography | performed 1 day before and 1 month after treatment
  Diffusion tensor imaging (DTI) is based on determining tissue structure by measuring diffusion rate and direction of movement of water molecules in vivo. DTI is the only in vivo method of mapping white-matter pathways in the human brain. Tractography is the technique for mapping white-matter structure with DTI data
Change in Fugl-Meyer Assessment Scale score(FMA) | performed 1 day before the end of the second week of the treatment and 1 day after the completion of the treatment
  FMA is a stroke-specific, performance-based impairment index. (0 point : Flaccid paralysis 100points=Normal).

IPD SHARING:
Plan to Share IPD: No
I do not to want to share IPD of my study. But if a researcher reaches me about the subject and wants me to share bended, I share IPD.